CLINICAL TRIAL: NCT07202234
Title: A Randomized Controlled Trial of Bacteriophage Cocktail Therapy for Multidrug-Resistant Gram-Negative Ventilator-Associated Pneumonia
Brief Title: Bacteriophage Cocktail Therapy for Multidrug-Resistant Gram-Negative Ventilator-Associated Pneumonia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Peking University Third Hospital (Other); Zhengzhou Central Hospital (Other); Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); The 8th medical center of chinese PLA general hospital (Unknown); The First Medical Center of Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, wang kaifei, Clinical Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Phage-2025YFC3408504
Record Dates: First submitted 2025-08-26; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: VAP - Ventilator Associated Pneumonia
Keywords: phage therapy; ventilator-associated pneumonia; phage cocktail
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): Nebulized normal saline inhalation therapy
  Interventions: Drug: Nebulized normal saline inhalation therapy
- phage therapy group (Experimental): Phage cocktail administered via nebulization
  Interventions: Drug: Phage cocktail administered via nebulization

INTERVENTIONS:
Drug: Phage cocktail administered via nebulization — Phage cocktail administered via nebulization，BID
  Arms: phage therapy group
Drug: Nebulized normal saline inhalation therapy — Nebulized normal saline inhalation therapy, BID
  Arms: control group

SUMMARY:
The purpose of this study is to systematically evaluate the efficacy and safety of bacteriophage cocktail therapy in patients with ventilator-associated pneumonia caused by Gram-negative bacterial infections.

DETAILED DESCRIPTION:
This study investigates the clinical application of bacteriophage therapy in severe infections through a prospective, randomized, multi-center trial targeting ventilator-associated pneumonia (VAP) caused by multidrug-resistant Gram-negative bacteria. The trial will comprehensively assess the efficacy, safety, and applicability of inhaled bacteriophage cocktail therapy, providing high-quality clinical evidence to support the establishment of an evidence-based framework for phage therapy. The primary endpoint is clinical response rate, with secondary endpoints including bacterial clearance and 28-day mortality, aiming to determine the therapeutic potential and clinical value of phage cocktails in VAP treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with ventilator-associated pneumonia (VAP);
2. Identified infection with MDR Klebsiella pneumoniae, Acinetobacter baumannii, or Pseudomonas aeruginosa via MROSE evaluation and antimicrobial susceptibility testing (AST) from this or other tertiary hospitals;
3. Aged 18 to 85 years;
4. Written informed consent obtained from the patient or legal guardian.

Exclusion Criteria:

1. Pregnant or breastfeeding women;
2. FiO₂ ≥ 70% or PEEP ≥ 15 cmH₂O;
3. Hemodynamic instability (vasopressor dose increased by ≥30% in the last 6 hours or norepinephrine > 0.5 μg/kg/min);
4. Known allergy to phage components.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate | From enrollment to the end of treatment (within 10 days of enrollment)

SECONDARY OUTCOMES:
Bacterial clearance rate | 10 days after enrollment
28-day mortality | 28 days after enrollment
Length of hospital stay | 28 days after enrollment
Length of invasive mechanical ventilation | 28 days after enrollment
CPIS score | 1，5，10 days after enrollment
  Full Title: Clinical Pulmonary Infection Score (CPIS);Range: Minimum: 0, Maximum: 12
  ;Interpretation: Higher score indicates more severe infection.
SOFA score | 1，5，10 days after enrollment
  Full Title: Sequential Organ Failure Assessment (SOFA) Score;Range: Minimum: 0, Maximum: 24
  ;Interpretation: Higher score indicates greater organ dysfunction.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT07202234/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-25): https://cdn.clinicaltrials.gov/large-docs/34/NCT07202234/ICF_001.pdf